CLINICAL TRIAL: NCT05713747
Title: A Multi-case Feasibility Study for "Life Skills Boot Camp": Mastering the Skills for Professional and Personal Success' Training Program
Brief Title: Life Skills Boot Camp Study (LEVELUP2)
Acronym: LEVELUP2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cyprus (Other)
Collaborators: VU University of Amsterdam (Other); University of Crete (Other); University of Jaén (Other)
Responsible Party: Principal Investigator, Prof. Georgia Panayiotou, Dr. Georgia Panayiotou, Professor of Clinical Psychology, Department of Psychology and Center for Applied Neuroscience, Principal Investigator, University of Cyprus
Other Study IDs: LEVELUP_Feasibility2
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Mental Health
Keywords: Emotion regulation
MeSH Terms: conditions — Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Life Skills Boot Camp — The boot camp is designed to be taken by undergraduate students across all disciplines with no pre-requisite coursework and students who participated in the "Life skills 101" course and have selected to participate in a boot camp training as part of their Individual Self Development Plan. The boot camp will consist of 3 training programs with 4 sessions (1.5 hour per session) each, including an introductory and a closing part.
  Content The boot camp was designed by a team of academics having several years of experience in clinical psychology, educational psychology, and health psychology. The focus of the bootcamp is to teach students practical skills in three different domains of soft skills: a) Interpersonal Skills, b) Resilience and Flexibility and c) Emotion Regulation.

SUMMARY:
In the present study, the investigators aim to examine a) the acceptability and feasibility of the "Life Skills Boot Camp", a series of soft skills trainings for students in higher education.

The acceptability and feasibility will be explored from the perspective of stakeholders, including students participating in trainings and trainers who provide them; b) to evaluate potential effectiveness of the training by measuring students' acquired knowledge and improvement on self-insight.

DETAILED DESCRIPTION:
The role of Higher Education in sustained economic growth, and social progress is critical. HE institutions (HEIs) as key 'future shaper' settings, host a significant proportion of talented youth, future workforce, and leader (Cawood, Dooris, & Powell, 2010; Suárez-Reyes, Muñoz Serrano, & Van den Broucke, 2019). Entering university marks a turning point for youth, since HEIs can empower young people to transform and expand skills to manage complex and global environmental and societal challenges.

Soft skills, such as the ability to set goals and achieve them, to regulate emotions, to demonstrate agility and adaptability, and manage interpersonal relationships, are now an emerging trend for tackling global economic and societal challenges (World Economic Forum, 2016; Organisation for Economic Co-operation and Development, 2019). In addition, soft skills related to mental and physical health, wellbeing and adjustment, have received growing interest over recent years, and have become even more critical in the context of emerging needs to build resilience in the face of the Covid-19 pandemic and in preparation for future crises (Bauer, et al. 2021; Liang, et al. 2020; Nearchou, et al. 2020; Rousseau, & Miconi, 2020).

Despite soft skills importance, evidence confirm a "skills gap", meaning that youth lack soft skills that are highly important in the workplace (Noah, & Aziz, 2020). Although students in HE commonly graduate with excellent technical academic skills to do well in their future profession, it is highly debated whether higher education graduates also have developed sufficient soft skills essential to do well at the workplace (Noah, & Aziz, 2020).

Given these challenges to individuals' academic performance, work achievement, and mental health, it would be advisable to equip students with the resources required for life success. As these skills become increasingly of central interest to communities, it becomes a pertinent question on how to expand them within the academic context by learning relevant information and practicing skills in a way that is responsive to the needs of the wider student community.

To deal with these situations, different types of skill training interventions/ competence-based education within HE, have been created to help students develop skills for self- development (e.g. Rubens et al., 2018) and alleviation of mental health symptoms/mental health promotion (for metanalyses see Conley, Durlak, & Kirsch, 2015; Conley et al., 2017; Yusufov et al., 2019). Current findings suggest that a) incorporating specific components (such as coping skills training or CBT and relaxation techniques for stress management, Yusufov et al., 2019) and b) specific training methodologies such as supervised skill training (Conley, Durlak, & Kirsch, 2015) or short-term/ brief trainings (Yusufov et al., 2019) may be beneficial for students and increase the feasibility of integrating these interventions in the HE context.

In addition to determining the active ingredients of interventions, defining pragmatic challenges, such as the best methodologies to coordinate and integrate such interventions within the HE context are also of key importance (Conley et al., 2017). Continued research is needed to identify the specific systems and practices that will place students in an active role to define self-development goals and practice, in a systematic and guided form, some of these soft skills in real life settings.

During the last decades, increasing attention toward multitiered frameworks of interventions has emerged, as an approach that takes into account the role of the context and the level of provided support to facilitate the personal competencies of all students (Jimerson, Burns, & VanDerHeyden, 2015; Arora et al. 2019). Τhe EU funded project LEVEL-UP (Ref: 2020-1-CY01-KA203-065985) is based on this kind of logic and aims to develop an innovative framework that lies in a 3- level support system that follows a linear, progressive fashion, starting from the broader application to the narrower one. According to the conceptualization of the project, in level 1, students will have the opportunity to gain up-to-date scientific knowledge on transversal skills through an introductory course. Through this course, students will be able to self-reflect on these skills and develop an Individual Skills Development Plan (ISDP). After completing the introductory course, each student will have the opportunity to broaden as well as to deepen specific transversal skills (based on their ISDP), through stepwise, guided and multi-contextual practical training. Specifically, students will be able to enroll in skills development programs (group-based) offered by experts within the HEI (level 2), practice, apply and refine them through feedback. Finally, in level 3, participants of level 2, who are identified through self- and instructor evaluation as presenting significant challenges in specific skills domains, would be able to develop and consolidate these skills under a more intensive and individualized supportive program.

The present study is part of LEVEL UP project and its focus is to test the conjunction of the two levels of the proposed framework: at level 1 students get research-informed knowledge on soft skills and self-reflect on the level of mastery of these skills, and at level 2 they develop specific skills through the participation in an intensive and supervised skills training. The primary goal of this study is to determine the feasibility both of delivering level 2 as a standalone low-intensity skills training (with no pre-requisite) and as a part of the two-level system (level 1 as a pre-requisite for to participate in level 2). Specifically, we aim to examine the feasibility and acceptability of embedding a series of group-based soft skills trainings within university educational operations. These trainings cover three vital soft skills training topics: a) how to regulate emotions, b) how to interact with others in an effective manner and c) ways to build flexibility and their resiliency.

Study aims/Objectives

The objective of this study is to assess the acceptability and feasibility of the "Life Skills Boot Camp", a series of soft skills trainings for students in higher education. The acceptability and feasibility will be explored from the perspective of stakeholders, including students participating in trainings and trainers who provide them. The specific objectives of the study are to:

1. Determine feasibility and acceptability of the skills training by

   1. estimating feasible recruitment and refusal rates.
   2. measuring key outcome domains such as completion rates, missing data, students-reported measures of social satisfaction.
   3. determining the acceptability of course resources and factors influencing this.
   4. measuring participants' willingness to participate in highly specialized soft skills training.
   5. determining the acceptability of the boot camps as standalone training.
2. Identify under which conditions the "Life skills boot camp" are of added value to students' personal and professional development by

   a. recording the antecedents associated to students' perceived usefulness of boot camps trainings. In specific, perspectives of both students with previous relevant experience (having a boot camps training as a follow up to a previous introductory soft skills course) and students with no relevant experience will be evaluated in terms of training usefulness.
3. Evaluate the preliminary changes in soft skills and mental health of HE students after implementing the two-level soft skills intervention.

   1. Examining changes in positive mental health, depression, anxiety and stress before the introductory course (level 1) and after the soft skills bootcamps (level 2) (only NL).
   2. Analysing changes in social, emotion regulation, coping and resilience skills before and after the soft skills bootcamps (level 2) (only NL).

ELIGIBILITY:
Inclusion Criteria:

* People who are enrolled as students in one of the four universities.

Exclusion Criteria:

* No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students from one of the following universities: University of Cyprus, Vrije Universiteit Amsterdam, Panepistimio Kritis and Universidad de Jaén, who will be enrolled in soft skills training. Participation in the research procedures will be voluntarily open to all students in the sample.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the program | up to 10 weeks
  At post-intervention, principal researchers involved in the development and delivery of the intervention in each site, will complete Structured Assessment of FEasibility (SAFE; Bird et al. 2014), a standardised measure of the feasibility of complex interventions (Bird et al. 2014). The SAFE measure comprises 16 items grouped into two sub-scales: Blocks (8 items) and Enablers (8 items). SAFE guidelines recommend that reviewers attend to the individual items of the scale, instead of using summary scores, since items have unequal weight.Τhe tool has shown excellent interrater reliability (k = 0.84, 95% CI 0.79-0.89) and test-retest reliability (k = 0.89, 95% CI 0.85-0.93).
Acceptability | up to 10 weeks
  At post-intervention, all participants will complete a course satisfaction/acceptability questionnaire. The questionnaire will consist of two parts: In part A (quantitative) students will be asked several Likert-scale questions, while part B (qualitative) while contain open-ended response questions relating to their experience, satisfaction, and the challenges/enablers associated with design and implementation of the course. Qualitative data from open-ended questions will be considered alongside the quantitative measures to assess the feasibility of the intervention. The feasibility and acceptability of the intervention will be evaluated, using multiple primary endpoints such as:
  1. Adherence (Total registrations, Attendance Rates, Homework Adherence, Dropouts, App Downloads, App use)
  2. Acceptability (Course acceptability, course satisfaction, perceptions measured by both Likert Scale Questionnaire and open-ended questions).
Instructors' perspectives | up to 10 weeks
  A brief post-questionnaire consisted of open-ended questions will explore instructors' experiences in terms of delivery of learning content and practical challenges faced during trainings.

SECONDARY OUTCOMES:
Emotion regulation skills | up to 10 weeks
  Difficulties with Emotion regulation Scale (DERS-18; Victor, & Klonsky, 2016) consists of 18-items on a 5- point Likert scale (1 'never' to 5 'almost always') measuring emotion regulation problems. It measures six subscales: (1) Nonacceptance of emotional responses; (2) difficulty engaging in goal-directed behavior, (3) impulse control difficulties; (4) lack of emotional awareness, (5) limited access to emotion regulation strategies; and (6) lack of emotional clarity. Total internal reliability is excellent: Cronbach's α = .91; subscales internal consistency is good to excellent: Cronbach's α = .77 to .9.
Coping and resilience skills | up to 10 weeks
  The Connor-Davidson Resilience Scale (CD-RISC-10; Connor, & Davidson, 2003) measures resilience on a 5-point Liker scale (1 'not true at all'to 5 'true nearly all the time'). Internal consistency is good (Cronbach's α = .87).
Perceived stress | up to 10 weeks
  Perceived stress scale (PSS-10; Cohen, Kamarck, & Mermelstein, 1983) consists of 10-items measuring stress levels on a 4- point Likert scale (0 'never' to 4 'very often'). Internal consistency is good (Cronbach's α = .84 to .86)
Interpersonal skills | up to 10 weeks
  Interpersonal Competence Questionnaire (brief form - ICQ-15; Coroiu, et al. 2014) consists of 1-items on a 5-point Liker scale (1 'I am always poor at this to 5 'I am expremely good at this) measuring interpersonal skills. It measures: (1) initiation; (2) Negative assertion; (3) Emotional support; (4) Disclosure; and (5) conflict management. Internal consistency is good (Cronbach's α = .87).
Positive mental health | up to 10 weeks
  Mental health Continuum-Short Form (MHC-SF; Keyes, 2006) consists of 14-items on a 6- point Likert scale (0 'never' to 5 'everyday'). It measures (1) emotional wellbeing (happiness, interest, satisfaction); (2) psychological wellbeing (selfacceptance, mastery, positive relations, personal growth, autonomy, purpose in life), and (3) social wellbeing (social contribution, integration, actualization, acceptance, coherence). Higher scores indicate greater levels of positive wellbeing.
  The instrument has shown good internal reliability for the total score (Cronbach's α = .89) and acceptable to good internal consistency for its subscales (Cronbach's α = .74 to 83).
Depression, anxiety and stress | up to 10 weeks
  Depression Anxiety Stress Scales (DASS-21;Henry, & Crawford, 2005) consist of three scales (7 items per scale) measuring states of depression, anxiety and stress on a 4 point Likert scale (0 'almost always' to 4 'never'). higher scores indicating a greater number of symptoms. The DASS-21 subscales show good internal consistency (Cronbach's α = 0.81- 0.88).

CONTACTS AND LOCATIONS:
Locations (4):
- University of Cyprus, Nicosia, Cyprus
- University of Crete, Rethymno, Greece
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands
- Universidad de Jaén, Jaén, Spain

IPD SHARING:
Plan to Share IPD: Undecided